CLINICAL TRIAL: NCT06572917
Title: Single-dose Prophylactic INdomethacin in Extremely Preterm Infants - A Multicenter Randomized Blinded Placebo-Controlled Trial (the SPIN RCT)
Brief Title: Single-dose Prophylactic INdomethacin in Extremely Preterm Infants
Acronym: SPIN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Souvik Mitra, MD PhD, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H24-02525
Record Dates: First submitted 2024-08-19; First posted 2024-08-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Extreme Prematurity; Intraventricular Hemorrhage; Morbidity;Newborn
Keywords: extremely preterm; severe intraventricular hemorrhage; mortality; prophylactic indomethacin
MeSH Terms: interventions — Indomethacin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The indomethacin and placebo will be provided to the bedside nurse as per allocation using pre-filled syringes masked with a yellow tape (as reconstituted indomethacin has a slightly yellow tinge). All members of the medical team and outcome assessors will remain blinded to the allocation throughout the trial duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-dose prophylactic indomethacin - SPIN (Experimental): Infants randomized to the SPIN group will receive a single 0.1 mg/kg dose of intravenous indomethacin within 12h of birth as a slow infusion over 20 mins.
  Interventions: Drug: Indomethacin
- Control (Placebo Comparator): Equal volume saline placebo administered intravenously over 20 mins
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indomethacin — Single dose of 0.1 mg/kg dose intravenous indomethacin as a slow infusion over 20 mins
  Other Names: Indocid
  Arms: Single-dose prophylactic indomethacin - SPIN
Drug: Placebo — Single dose of intravenous normal saline placebo as a slow infusion over 20 mins
  Other Names: Normal saline
  Arms: Control

SUMMARY:
In Canada, about 900 babies each year are born very early (<26 weeks of gestation) and have a high chance of dying or having a serious bleed in the brain. Families of these extremely preterm babies consider preventing severe brain bleeding as critical to their child's health and well-being. A medicine called indomethacin, when given intravenously in 3-doses, is known to reduce severe brain bleeding. But use of this drug is variable among clinicians working in the neonatal intensive care unit (NICU) due to (a) its side effects on the gut; (b) possible harm when used with other medications; (c) a notion that despite reducing brain bleeds, the child's long-term brain development is not improved. Emerging evidence suggests that a single low-dose indomethacin regimen may be equally effective in reducing severe brain bleeding as compared to a traditional 3-dose regimen.

The investigators propose a blinded randomized controlled trial, a study design where babies born <26 weeks will be randomly assigned within 12 hours of birth to either a single dose of intravenous indomethacin or similar looking placebo in the form a saline solution. The study will test if a single dose indomethacin regimen is effective in improving survival of these babies without the devastating complication of severe brain bleeding. In this study the care providers and researchers will be unaware as to which baby receives indomethacin and which baby receives placebo to ensure no one's expectations or biases can influence the results.

The investigators will conduct the study in multiple NICUs across Canada, the United States and Australia in 2 phases: First, an internal pilot phase that will enroll 104 babies born <26 weeks or <750 g birth weight over a period of 1 year. If the investigators are successful in achieving their target enrolment in the pilot phase, they will move on to the second phase and continue enrollment up to a total of 500 babies born <26 weeks or <750 g birth weight over a period of 3 years. The total of 500 babies will include the 104 babies enrolled in the first phase of the study. This study will help the investigators determine in the most unbiased way whether a single dose of indomethacin given immediately after birth in the smallest babies born <26 weeks of gestation can safely and effectively reduce severe brain bleeding.

DETAILED DESCRIPTION:
BACKGROUND & IMPORTANCE In Canada, about 900 infants are born extremely preterm at <26 weeks of gestation (GA); nearly four out of 10 of them do not survive or develop severe intraventricular hemorrhage (sIVH). Existing evidence shows that a 3-dose regimen of prophylactic intravenous indomethacin (0.1mg/kg/dose every 24h for 3 doses most commonly used clinically) results in a significant reduction in sIVH, an outcome deemed critical by families. However, use of the conventional 3-dose regimen has declined among clinicians due to perceived adverse effects on the gut, presumed lack of long-term neurodevelopmental benefit and preclusion of other early therapeutic interventions such as ibuprofen or hydrocortisone due to potential increased risk of gut perforation with concomitant use with indomethacin.

Recent pharmacokinetic studies show that indomethacin drug clearance is significantly reduced in infants born ≤26 weeks GA in the first week of life due to their developmental immaturity; and consequently a single 0.1 mg/kg dose likely maintains therapeutic levels for at least 72h - the most critical period of sIVH onset in these smallest infants. However, no RCTs have yet been conducted to establish effectiveness and safety of this single dose regimen in this highest risk population.

GOAL(S) / RESEARCH AIMS Primary goal: To determine the effectiveness and safety of single dose prophylactic indomethacin to prevent morbidity and mortality in extremely preterm infants born <26 weeks GA.

The investigators hypothesize that in preterm infants born <26 weeks GA, when compared to placebo, a single 0.1 mg/kg dose of intravenous indomethacin given prophylactically within the first 12 hours of birth will improve survival without sIVH.

METHODS/APPROACHES/EXPERTISE Study design: Multicenter, blinded, placebo-controlled, individually randomized, Bayesian design RCT Population: Preterm infants born <26 weeks GA and/or <750 g birth weight Intervention: Prophylactic indomethacin: Single-dose intravenous indomethacin (0.1 mg/kg) given within 12 hours of birth. Comparison: Equal volume saline placebo.

Sample size and analysis: The proposed sample size is 500 neonates (250 per arm). The primary analysis will utilize a Bayesian approach using an informative prior that assumes a 5% expected net benefit (in absolute risk difference) with an uncertainty of 5%, with regards to the primary outcome. The trial will be considered successful if it shows that the posterior probability of a positive net benefit is at least 90%.

Setting: Neonatal intensive care units across Canada, the United States and Australia over 3 years. The study will be conducted in 2 phases: (i) an internal pilot phase that will enroll 104 infants born <26 weeks or <750 g birth weight over a period of 1 year; (ii) If the investigators are successful in achieving their target enrolment in the pilot phase, they will move on to the second phase and continue enrollment up to a total of 500 infants born <26 weeks or <750 g birth weight over a period of 3 years. The total of 500 infants will include the 104 infants enrolled in the first phase of the study.

Primary outcome: Survival without sIVH (grades 3 and 4) at hospital discharge Secondary outcomes include in-hospital clinical outcomes; white matter injury on MRI at term corrected age; neurodevelopmental impairment at 24 (±6) months; pharmacokinetic (PK) profile of single-dose indomethacin; total hospital costs and costs per sIVH or death averted.

EXPECTED OUTCOMES This will be the first RCT to explore the effectiveness and safety of single dose prophylactic indomethacin exclusively in infants born <26 weeks GA who are at the highest risk of severe IVH and death. Apart from the primary and secondary clinical outcomes, this trial will describe the PK profile of single dose indomethacin to establish the ideal therapeutic window for sIVH prevention as well as ascertain the value for money of this therapy in preventing death and sIVH in infants born <26 weeks GA.

ELIGIBILITY:
Inclusion Criteria:

* Extremely preterm infants born <26 completed weeks of GA and/or extremely low BW infants born <750g

Exclusion Criteria:

* antenatal diagnosis of duct dependent CHD
* acute hypoxic respiratory failure [defined as fraction of inspired oxygen (FiO2)>0.60 for ≥2h)
* inhaled nitric oxide (iNO) therapy due to suspected or confirmed acute pulmonary hypertension (PH)
* receipt of prophylactic or therapeutic hydrocortisone
* antenatal diagnosis of renal anomalies
* initial platelet count <50x109/L
* decision to withhold/withdraw life-sustaining treatments

Ages: 0 Hours to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Survival without severe intraventricular hemorrhage (sIVH) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Any IVH more than grade 2 (i.e., grade 3, grade 4/intraparenchymal hemorrhage/perventricular hemorrhagic infarction is classified as sIVH

SECONDARY OUTCOMES:
Mortality | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Severe IVH | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Any IVH more than grade 2 (i.e., grade 3, grade 4/intraparenchymal hemorrhage/perventricular hemorrhagic infarction is classified as sIVH
Gastrointestinal perforation | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Necrotizing enterocolitis (NEC) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Bell Stage ≥stage 2
Acute kidney injury (AKI) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Defined as ≥stage 1 according to the Neonatal AKI KDIGO classification)
Persistent patent ductus arteriosus | 7 days postnatal age
  Defined as presence of PDA status on day 7 echocardiogram
Procedural PDA closure | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Definitive PDA closure either by surgical ligation or interventional percutaneous catheter based closure
Chronic pulmonary hypertension | birth through 36 weeks' postmenstrual age (PMA)
  Echocardiographic evidence of chronic pulmonary hypertension
Grade 3 Bronchopulmonary dysplasia (BPD) | birth through 36 weeks' postmenstrual age (PMA)
  Defined as need for invasive mechanical ventilation at 36 weeks' postmenstrual age
Pulmonary hemorrhage | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Defined as blood stained respiratory secretions with an acute significant increase in respiratory requirements (Mean Airway Pressure>12 cm H2O and/or Fraction of inspired O2>60%
Duration of invasive mechanical ventilation in days | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Postnatal corticosteroid use | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
IVH (any grade) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Periventricular leukomalacia (any grade) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
White matter injury (WMI) | Term corrected age (approximately 20 weeks postnatal age)
  Defined on MRI brain as discrete areas of abnormal white matter T1 hyperintensity in the absence of marked T2 hypo-intensity, or by low-intensity T1 foci
Severe retinopathy of prematurity (ROP) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Defined as ROP ≥stage 3
Major neurodevelopmental impairment | 24 (±6) months postmenstrual age (PMA)
  Defined as any one of: (i) CP with an inability to walk unassisted; (ii) major developmental delay involving cognition or language or (iii) visual (cannot fixate/legally blind, or corrected acuity <6/60 in both eyes), or hearing impairment (requiring a hearing aid or cochlear implants)

OTHER OUTCOMES:
Pharmacokinetic outcomes | 7 days postnatal age
  clearance, volume of distribution and plasma exposure of single-dose indomethacin
Health Economic outcomes | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Total healthcare costs (measured to first discharge home); cost per sIVH or death averted; and cost per death averted
Primary feasibility outcomes (during the internal pilot) | Through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  (1) Proportion of eligible infants randomized during the internal pilot; (2) Proportion of randomized infants with no reported protocol deviation during the internal pilot
Secondary feasibility outcomes (during the internal pilot) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  (1) Reasons for non-recruitment and non-adherence to protocol; (2) qualitative views of parents and neonatologists on recruitment strategies

CONTACTS AND LOCATIONS:
Overall Officials: Souvik Mitra, MD, PhD, Principal Investigator — University of British Columbia
Locations (15):
- United States (5):
  - Kaiser Roseville, Roseville, California
  - UC Davis Health, Sacramento, California
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Texas Health Harris Methodist Hospital Fort Worth, Fort Worth, Texas
  - Welcome to Baylor Scott & White Health, Fort Worth, Texas
- Australia (2):
  - Mercy Hospital for Women, Melbourne, Victoria
  - Monash Children's Hospital, Melbourne, Victoria
- Canada (8):
  - Foothills Medical Center & Alberta Children's Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - BC Women's Hospital, Vancouver, British Columbia
  - IWK Health, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data on clinical outcomes collected during the trial will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon as possible, wherever legally and ethically possible. In addition, data from the trial will be made available upon reasonable request.